CLINICAL TRIAL: NCT04665609
Title: Safety and Effectiveness of Thermal Ablation Combined With Anlotinib and TQB2450 Solution for Advanced Hepatocelualr Carcinoma
Brief Title: Thermal Ablation Combined With Anlotinib and TQB2450 Solution for HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 301jrcsk-lp-yj
Record Dates: First submitted 2020-11-30; First posted 2020-12-11 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Carcinoma; Thermal Ablation; Anlotinib; PDL-1
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib and TQB2450 solution (Experimental): Microwave ablation will be performed according to patients' tumor number, size and liver function. Oral anlotinib (12 mg/d) will be administered and its cycle is defined as 2 weeks on-treatment followed by 1 week off-treatment. Patients will be given 1200 mg TQB245 solution intravenously every 3 weeks. The treatment continues until disease progression or treatment intolerance. Anlotinib and TQB2450 solution will be given after 2 weeks of microwave ablation procedure.
  Interventions: Drug: Anlotinib and TQB2450 solution
- TQB2450 Solution (Active Comparator): Microwave ablation will be performed according to patients' tumor number, size and liver function. Patients will be given 1200 mg TQB245 solution intravenously every 3 weeks.TQB2450 solution will be given after 2 weeks of microwave ablation procedure.
  Interventions: Drug: TQB2450 solution

INTERVENTIONS:
Drug: Anlotinib and TQB2450 solution — Anlotinib is a novel multitarget tyrosine kinase inhibitor, inhibiting tumour angiogenesis and proliferative signalling. TQB2450 solution is a new novel of PD-L1 inhibitor made by Crown Bioscience and CHIATAI TIANQING(CTTQ PHARMA).
  Arms: Anlotinib and TQB2450 solution
Drug: TQB2450 solution — TQB2450 solution is a new novel of PD-L1 inhibitor made by Crown Bioscience and CHIATAI TIANQING(CTTQ PHARMA).
  Arms: TQB2450 Solution

SUMMARY:
In this study, investigators aimed to evaluated the efficacy and safety of microwave ablation combined with anlotinib and TQB2450 Solution in patients with advanced hepatocellular carcinoma. Patients were randomly assigned at a one-to-one ratio to receive microwave ablation plus anlotinib and TQB2450 Solution or microwave ablation plus TQB2450 Solution. Primary end points were objective response rate(ORR). Second end points include overall survival, progression-free survival and disease control rate. Safety was assessed in all patients.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG PS score: 0-1, Life expectancy of 3 months or more
2. Subjects must have confirmed diagnosis of HCC
3. BCLC B and C grade
4. At least 1 measurable target lesion according to mRECIST
5. Child-Pugh score A to B
6. No locoregional therapy within 4 weeks before enrollment for patients with unresectable HCC or tumor progression after locoregional therapy; All toxicities related to prior treatments must be resolved to Grade ≤1
7. No prior treatment with anti-angiogenic drugs or any anti-PD-1 agent within 4 weeks before enrollment
8. HBV DNA<500IU/mL
9. Adequate organ function within 14 days before enrollment
10. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to the start of study drug. Women must not be breastfeeding. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment
11. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol

Exclusion Criteria:

1. Prior liver transplant
2. Any prior (within 1 year) or current clinically significant ascites as measured by physical examination and that requires active paracentesis for control
3. Prior treatment with an anti-PD-L1
4. Active autoimmune disease that has required systemic treatment in past 2 years
5. Known or suspected allergy to Anlotinib and TQB2450 Solution or study drug components；History of severe hypersensitivity reaction to any monoclonal antibody
6. Has received a live-virus vaccination within 30 days of planned treatment start.
7. Subjects with CNS metastases are not eligible, unless they have completed local therapy (eg, whole brain radiation therapy [WBRT], surgery or radiosurgery) and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs (eg, radiologic) or symptoms of brain metastases must be stable for at least 4 weeks before starting study treatment
8. Subjects with any active, known, or suspected autoimmune disease； Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
9. HBV DNA ≥ 1000 IU/ml，HCV RNA
10. New York Heart Association congestive heart failure of grade II or above, unstable angina, myocardial infarction within the past 6 months, or serious cardiac arrhythmia associated with significant cardiovascular impairment within the past 6 months, Prolongation of QTc (Fridericia formula) interval to >480 ms
11. Dysfunction of blood coagulation （INR>1.5 or APTT>1.5×ULN）, Bleeding or thrombotic disorders
12. Anticoagulants requiring therapeutic INR monitoring, eg, warfarin or similar agents. Antiplatelet agents and low molecular weight heparin are prohibited throughout the study
13. Active infection (any infection requiring systemic treatment)
14. History of solid organ or hematologic transplant
15. Any medical or other condition which, in the opinion of the investigator, would preclude participation in a clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-05 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 2-year
  Objective Response Rate

SECONDARY OUTCOMES:
OS | 2-year
  Overall Survival
PFS | 2-year
  Progression-free Survival
DCR | 2-year
  Disease Control Rate
EORTC QLQ C30 | Change from baseline health related quality of life at 2 years
  Impact of treatment on Health Related Quality of Life (HRQoL) for subjects treated using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire. EORTC QLQ C30 scales were grouped and converted to score 0 to 100 according to the scoring manual; a higher score represents a more severe symptom or problem.
EORTC QLQ-HCC18 | Change from baseline health related quality of life at 2 years
  Impact of treatment on Health Related Quality of Life (HRQoL) for subjects treated using HCC-specific EORTC QLQ-HCC18 questionnaire. EORTC QLQ-HCC18 scales were grouped and converted to score 0 to 100 according to the scoring manual; a higher score represents a more severe symptom or problem.
AE | 2-year
  Incidence of Adverse Events
SAEs | 2-year
  Incidence of Severe Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China